CLINICAL TRIAL: NCT06054958
Title: POTS-CFS Study: A Case-Control Study on Exertion and Orthostatic Intolerance in the Context of Pediatric ME/CFS
Brief Title: POTS-CFS Study: Orthostatic Intolerance in the Context of Pediatric ME/CFS
Acronym: POTS-CFS
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: University Hospital, Aachen (Other)
Responsible Party: Sponsor
Other Study IDs: POTS-CFS
Record Dates: First submitted 2023-08-16; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-07

CONDITIONS: Chronic Fatigue Syndrome in Adolescence; Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ME/CFS: ME/CFS: adolescents aged 14-17 years, fulfilling diagnostic criteria for ME/CFS according to Rowe e 2017, Jason 2006, CCC 2003, and/ or IOM 2015 at the time of recruitment.
  Methods: Semi-structured interview, questionnaires, passive 10-minute standing test (NASA lean test), blood sampling.
- Healthy Controls (HC): HC: adolescents aged 14-17, clinically healthy without any known underlying disease and with no prescription drugs (except contraception).
  Methods: Semi-structured interview, questionnaires, passive 10-minute standing test (NASA lean test), blood sampling.

SUMMARY:
Pilot-case-control study on exertion and orthostatic intolerance of adolescents with myalgic encephalomyelitis/ chronic fatigue syndrome (ME/CFS) compared to age-matched healthy controls (HC).

DETAILED DESCRIPTION:
ME/CFS is a complex disease. Symptoms include orthostatic intolerance (OI) such as postural tachycardia syndrome (PoTS). PoTS in ME/CFS can significantly impair everyday function and social participation. Yet, data in affected adolescents are rare and inconsistent.

This pilot-case-control study study aimed at characterizing OI in adolescents aged 14-17 years with ME/CFS and age-adapted HC, comparing the results with other clinical features of both such as exertion intolerance, fatigue, and health-related quality of life, and suggesting a standardized tool for diagnostics.

ME/CFS was diagnosed according to the Clinical Canadian Criteria (CCC 2003), criteria of the former Institute of Medicine (IOM 2015), the diagnostic work sheet developed by Rowe 2017, and/or the pediatric case suggested by Jason 2006. Questionnaires were used to evaluate symptoms (e.g. post-exertional malaise, fatigue, anxiety, depression), and health-related quality of life. A standardized specific interview was performed to assess the medical history of OI (HOI). Heart rate (HR) and blood pressure were evaluated every minute during a passive 10-min standing test (NASA lean test) in the morning with empty stomach and without morning medication.

Data were evaluated according to the PoTS criteria defined in 2019 at the National Institutes of Health Expert Consensus Meeting and by the International Classification of Diseases (ICD-11) (8D89.2). Frequency and type of OI, including PoTS, were examined in both groups and outcomes compared to parameters from questionnaires. Based on the results, novel standards for OI diagnostics were suggested.

ELIGIBILITY:
Inclusion Criteria:

1. Cases (ME/CFS):

   - ME/CFS diagnosed by the indicated clinical criteria
2. Healthy Controls

   * clinically healthy
   * no known underlying disease
   * no prescription medication (except contraception)

Exclusion Criteria:

* Any contraindication for NASA lean test (cardiac failure, severe aortic stenosis, inability to stand)
* pregnancy
* breastfeeding.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents with ME/CFS and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Heart Rate during Passive 10-min. standing test | one time point during study from study start until study completion, approximately 1 year
  Heart rate during Passive 10-Min. standing test (NASA lean test)
Blood Pressure during Passive 10-min. standing test | one time point during study from study start until study completion, approximately 1 year
  blood pressure, pulse pressure (calculated by systolic and diastolic blood pressure) during Passive 10-Min. standing test (NASA lean test)
Symptoms during Passive 10-Min. standing test | one time point during study from study start until study completion, approximately 1 year
  Symptoms during Passive 10-Min. standing test (NASA lean test): Yes/No
O2-Saturation during Passive 10-Min. standing test | one time point during study from study start until study completion, approximately 1 year
  O2-Saturation during Passive 10-Min. standing test (NASA lean test)
Presence of Orthostatic Intolerance: Semistructured Interview | one time point during study from study start until study completion, approximately 1 year
  Semistructured Interview, History of Orthostatic Intolerance (OI): Yes/No
Number of orthostatic Symptoms: Semistructured Interview | one time point during study from study start until study completion, approximately 1 year
  Semistructured Interview, Number of Symptoms
Number of participants with a diagnosis of PoTS, Orthostatic Intolerance and related diagnoses | one time point during study from study start until study completion, approximately 1 year
  History of OI and Nasa lean test together result in an orthostatic diagnosis, Fulfilling of PoTS-Criteria at study visit is evaluated
Presence of ME/CFS-specific Symptoms (Munich Berlin Symptom Questionnaire) | one time point during study from study start until study completion, approximately 1 year
  Questionnaire: number of relevant symptoms. Likert Scale "0-4" of severity and frequency for each symptom: A symptom is relevant with a severity and frequency of each at least "2" on the Likert Scale. Minimum: 0 relevant symptoms (best), Maximum: 60 relevant symptoms (worst).
Presence of Post-exertional malaise (DePaul Symptom Questionnaire -Post exertional Malaise: DSQ-PEM) | one time point during study from study start until study completion, approximately 1 year
  Questionnaire, Binary Outcome: Post-exertional Malaise Yes/No
Self-estimated level of Quality of Life: EQ-5D-5L: Index | one time point during study from study start until study completion, approximately 1 year
  Questionnaire: Index (0 worst - 1 best)
Self-estimated level of Quality of Life: EQ-5D-5L: Visual Analog Scale | one time point during study from study start until study completion, approximately 1 year
  Visual Analog Scale (0 worst - 100 best)
Screening via Public Health Questionnaire-4 (PHQ-4) | one time point during study from study start until study completion, approximately 1 year
  Ultra-Short-4-item-Screening for Anxiety/Depression: Scale (0 Symptom occurs never - 3 Symptom occurs almost every day)
Malmö PoTS Score (MAPS) | one time point during study from study start until study completion, approximately 1 year
  Orthostatic Symptoms Severity, Scale (0 no symptom burden - 120 highest symptom burden)

SECONDARY OUTCOMES:
Levels of serum antibodies against EBV | one time point during study from study start until study completion, approximately 1 year
  Levels of Autoantibodies at study visit
Levels of serum antibodies against SARS-CoV-2 | one time point during study from study start until study completion, approximately 1 year
  Levels of autoantibodies at study visit
Levels of serum autoantibodies | one time point during study from study start until study completion, approximately 1 year
  Levels of autoantibodies at study visit

CONTACTS AND LOCATIONS:
Locations (1):
- MRI Chronic Fatigue Center for Young People (MCFC) Children's Hospital, Technical University of Munich & Munich Municipal Hospital Munich, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.pots-dysautonomia.net/symposium-2022
- See also: Related Info — https://www.pots-dysautonomia.net/studienteilnahme
- See also: Related Info — https://lost-voices-stiftung.org/forschungsfoerderung/